CLINICAL TRIAL: NCT00649584
Title: A Phase I Dose Escalation Study of Weekly SGN-35 Monotherapy and in Combination With Gemcitabine in Patients With Relapsed/Refractory CD30-positive Hematologic Malignancies
Brief Title: A Phase I Dose Escalation Study of SGN-35 Alone and in Combination With Gemcitabine for CD30-Positive Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision not to enroll cohorts of combined SGN-35 and gemcitabine therapy.
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG035-0002
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin
Keywords: Antigens, CD30; Antibody-Drug Conjugate; Antibodies, Monoclonal; monomethyl auristatin E; Combined Modality Therapy; Drug Therapy; Immunotherapy; Lymphoma, Non-Hodgkin; Disease, Hodgkin; Lymphoma, Large-Cell, Anaplastic; Hematologic Diseases; Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Non-Hodgkin; Hematologic Diseases; Lymphoma | interventions — Brentuximab Vedotin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SGN-35 alone or in combination with gemcitabine
  Interventions: Drug: SGN-35; Drug: gemcitabine

INTERVENTIONS:
Drug: SGN-35 — IV; 0.4 up to 1.8 mg/kg weekly 3 out of 4 weeks; minimum of two 28-day cycles
  Other Names: brentuximab vedotin
Drug: gemcitabine — IV; 1000 mg/m2 weekly 3 out of 4 weeks
  Other Names: Gemzar

SUMMARY:
This study will examine the safety profile of SGN-35 alone and in combination with gemcitabine. The study will test increasing doses of SGN-35 given weekly to small groups of patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD30-positive hematologic malignancy.
* Patients with HL must have failed systemic chemotherapy.
* Patients with other CD30-positive malignancies (including ALCL) must be beyond first remission or refractory to front line chemotherapy.
* Patients must have measurable disease of at least 1.5 cm as documented by radiographic technique.

Exclusion Criteria:

* Current diagnosis of primary cutaneous ALCL (systemic ALCL eligible).
* History of allogeneic stem cell transplant.
* Patients who have had previous treatment with any anti-CD30 antibody.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and laboratory abnormalities | 1 month after last dose

SECONDARY OUTCOMES:
PK profile | 2 months after last dose
Immunogenicity (anti-SGN-35 antibodies) | 1 month after last dose
Anti-tumor activity | 1 month after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Dana Kennedy, PharmD, Study Director — Seagen Inc.
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University Medical Center, Palo Alto, California
  - University of Miami, Miami, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Fanale MA, Forero-Torres A, Rosenblatt JD, Advani RH, Franklin AR, Kennedy DA, Han TH, Sievers EL, Bartlett NL. A phase I weekly dosing study of brentuximab vedotin in patients with relapsed/refractory CD30-positive hematologic malignancies. Clin Cancer Res. 2012 Jan 1;18(1):248-55. doi: 10.1158/1078-0432.CCR-11-1425. Epub 2011 Nov 11. PMID 22080439